CLINICAL TRIAL: NCT01755403
Title: Population Pharmacokinetics in Benznidazole-treated Adults With Chronic Chagas Disease. Benznidazole Pharmacokinetics and Adverse Reactions Relationship.
Brief Title: Population Pharmacokinetics in Benznidazole-treated Adults With Chronic With Chagas Disease
Acronym: CINEBENZ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barcelona Centre for International Health Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINEBENZ
Record Dates: First submitted 2012-12-19; First posted 2012-12-24 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Chagas Disease
MeSH Terms: conditions — Chagas Disease | interventions — benzonidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Benznidazole (Other)
  Interventions: Drug: Benznidazole

INTERVENTIONS:
Drug: Benznidazole

SUMMARY:
o study population pharmacokinetics in Benznidazole-treated adult patients with Chronic Chagas Disease to get information to optimize drug doses.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Chronic Chagas Disease diagnosed by 2 different and positive serological tests.
* Patients with Chronic Chagas Disease who are going to start treatment with Benznidazole.
* Any gender.
* All the participants must agree to participate in the study and must sign the informed consent.

Exclusion Criteria:

* Patients younger than 18.
* Patients with previous hypersensitivity to Benznidazole.
* Immunocompromised patients as AIDS, cancer, chemotherapy, longterm corticoids need, primary immunodeficiency, or any other.
* Hepatic dysfunction
* Renal dysfunction: serum creatinin higher than 3 mg/dl.
* Pregnancy or lactation.
* Low adhesion to treatment or check-up.
* Impossibility of follow-up.
* Severe adverse reaction to Benznidazole.
* Any other situation that could be risky for the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Population pharmacokinetic parameters of Benznidazole | 2 months (treatment period)
  Population pharmacokinetic model development

SECONDARY OUTCOMES:
Adverse reactions | 2 months (treatment period)
  Number of participants with adverse events. Severity of adverse events. Relationship between adverse event and drug concentration.

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Gascón, PhD, Principal Investigator — Barcelona Centre for International Health Research (CRESIB)
Locations (1):
- International Health Department, Hospital Clinic, Barcelona, Barcelona, Catalonia, Spain

REFERENCES:
- [Derived] Aldasoro E, Posada E, Requena-Mendez A, Calvo-Cano A, Serret N, Casellas A, Sanz S, Soy D, Pinazo MJ, Gascon J. What to expect and when: benznidazole toxicity in chronic Chagas' disease treatment. J Antimicrob Chemother. 2018 Apr 1;73(4):1060-1067. doi: 10.1093/jac/dkx516. PMID 29351667
- [Derived] Soy D, Aldasoro E, Guerrero L, Posada E, Serret N, Mejia T, Urbina JA, Gascon J. Population pharmacokinetics of benznidazole in adult patients with Chagas disease. Antimicrob Agents Chemother. 2015;59(6):3342-9. doi: 10.1128/AAC.05018-14. Epub 2015 Mar 30. PMID 25824212